CLINICAL TRIAL: NCT00552357
Title: Clinical Risk Factors for Primary Graft Dysfunction
Brief Title: Risk Factors That Increase the Chance of Developing Primary Graft Dysfunction After Lung Transplantation
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Columbia University (Other); University of Alabama at Birmingham (Other); Vanderbilt University (Other); Stanford University (Other); Johns Hopkins University (Other); University of Michigan (Other); Duke University (Other); University of Pittsburgh (Other); University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 1417; R01HL087115-01A1 (NIH)
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Primary Graft Dysfunction; Lung Transplantation
MeSH Terms: conditions — Primary Graft Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Primary graft dysfunction (PGD) is a severe lung complication that can occur in the days after lung transplant surgery. This study will analyze blood samples to determine if high levels of certain chemicals may increase the risk of developing PGD after a lung transplant.

DETAILED DESCRIPTION:
PGD is a severe complication that affects up to 25% of lung transplant patients following surgery. Pulmonary edema, which is an abnormal build-up of fluid in the lungs, and hypoxemia, which is low blood oxygen levels, are two common symptoms that individuals with PGD experience. Treatment for PGD is often expensive, and it is the leading cause of death following lung transplantation. Many potential lung donors and recipients are considered unsuitable for lung transplantation because of concern for the development of PGD. Increased levels of chemicals that are involved in bleeding and clotting, including protein C, and certain markers of oxidant stress, which can cause damage to the body's cells and tissues, may increase a person's risk of developing complications following a lung transplant. The purpose of this study is to analyze blood samples to determine if elevated levels of certain chemicals may be associated with an increased risk of developing PGD after lung transplantation.

This study will enroll individuals who are undergoing lung or heart and lung transplantation. Blood samples will be collected from participants prior to surgery, immediately following surgery, and 24 hours after surgery. Study researchers will also review participants' medical records. There will be no additional study visits.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing lung or combined heart and lung transplantation

Exclusion Criteria:

* Undergoing combined organ transplantation other than heart and lung transplantation

Ages: 13 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People undergoing lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 1150 (Estimated)
Dates: Start 2007-12; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Primary graft dysfunction, defined by the ISHLT criteria | Measured within 72 hours following transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jason D. Christie, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Diamond JM, Cantu E, Calfee CS, Anderson MR, Clausen ES, Shashaty MGS, Courtwright AM, Kalman L, Oyster M, Crespo MM, Bermudez CA, Benvenuto L, Palmer SM, Snyder LD, Hartwig MG, Todd JL, Wille K, Hage C, McDyer JF, Merlo CA, Shah PD, Orens JB, Dhillon GS, Weinacker AB, Lama VN, Patel MG, Singer JP, Hsu J, Localio AR, Christie JD. The Impact of Donor Smoking on Primary Graft Dysfunction and Mortality after Lung Transplantation. Am J Respir Crit Care Med. 2024 Jan 1;209(1):91-100. doi: 10.1164/rccm.202303-0358OC. PMID 37734031
- [Derived] Diamond JM, Lee JC, Kawut SM, Shah RJ, Localio AR, Bellamy SL, Lederer DJ, Cantu E, Kohl BA, Lama VN, Bhorade SM, Crespo M, Demissie E, Sonett J, Wille K, Orens J, Shah AS, Weinacker A, Arcasoy S, Shah PD, Wilkes DS, Ware LB, Palmer SM, Christie JD; Lung Transplant Outcomes Group. Clinical risk factors for primary graft dysfunction after lung transplantation. Am J Respir Crit Care Med. 2013 Mar 1;187(5):527-34. doi: 10.1164/rccm.201210-1865OC. Epub 2013 Jan 10. PMID 23306540